CLINICAL TRIAL: NCT06825377
Title: Comparing the Effects of High-protein Nutritional Support with Standard Protein Nutritional Support Through the Administration of Whey Protein Supplements on Clinical Outcomes of Critically Ill Patients At Risk for Refeeding Syndrome: a Randomized Comparative Clinical Trial
Brief Title: Comparing High-protein Vs. Standard Protein Nutritional Support in Critically Ill Patients At Risk for Refeeding Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 450/1272
Record Dates: First submitted 2025-02-02; First posted 2025-02-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Malnutrition; Refeeding Syndrome; At Risk for Refeeding Syndrome
Keywords: Refeeding syndrome; Critically ill; High-protein; Complication; Malnutrition; mortality
MeSH Terms: conditions — Critical Illness; Malnutrition; Refeeding Syndrome | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-protein (Experimental): The target protein intake of 2 grams per kilogram of body weight per day will be gradually introduced, starting at a low level, through nutritional support, with whey protein powder added if needed as a supplement.
  Interventions: Dietary Supplement: Whey protein
- Standard-protein (Active Comparator): The target protein intake of 1.3 grams per kilogram of body weight per day will be gradually introduced, starting at a low level, through nutritional support, with whey protein powder added if needed as a supplement.
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Whey protein powder will be provided with nutritional support in both groups if needed to meet the target protein intake.

SUMMARY:
The goal of this clinical trial is to determine the optimal protein administration strategy for enhancing both nutritional and clinical outcomes, as well as reducing complications and mortality in ICU patients at risk for refeeding syndrome (RS). This study will include critically ill patients at risk for RS who are receiving supportive nutrition. The primary hypothesis is that higher protein intake will lead to a decreased incidence of refeeding syndrome. It is also expected that patients receiving more protein will have better clinical outcomes, lower mortality, and shorter ICU and hospital stays.

DETAILED DESCRIPTION:
Patients will be randomly assigned to two groups: the high-protein group and the standard-protein group. Upon ICU admission, and after meeting the inclusion criteria and identifying a risk of refeeding syndrome (RS), they will be allocated to one of the two groups. Patient selection for RS risk will be based on the diagnostic criteria outlined in the 2020 ASPEN guidelines. The m-NUTRIC and APACHE II scores will be calculated for all patients at ICU admission and 24 hours before the initiation of feeding. Monitoring for multi-organ dysfunction syndrome (MODS) will involve daily laboratory tests and organ failure assessment using the SOFA score.

Before starting the nutritional intervention, all patients will receive 100 mg of thiamine daily for one week, along with a daily multivitamin-mineral supplement. Due to the risk of RS, calorie intake will begin at low levels and will be cautiously increased in both groups. To calculate the energy needs, ideal body weight will be used. In the high-protein group, the target protein intake will be 2 grams per kilogram of body weight per day, while in the standard-protein group, it will be 1.3 grams per kilogram of body weight per day. Protein will be introduced gradually, starting from a low level, as part of nutritional support, with whey protein powder added if needed as a supplement. If serum creatinine levels rise, protein powder will be removed from the patient's diet. The intervention duration will be 14 days, with a minimum of 5 days.

The primary clinical outcome is the incidence of refeeding syndrome (RS), while secondary outcomes include the occurrence of infections, hospital length of stay, ICU length of stay, multi-organ failure, and mortality within 45 days of admission. RS will be diagnosed according to the 2020 ASPEN guidelines. Serum concentrations of potassium, magnesium, phosphate, glucose, urea, and creatinine will be measured daily for one week.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to cooperate and complete the informed consent form by the patient or legal guardian;
* age ≤ 18 years and < 65 years;
* Non-pregnant and non-lactating;
* Serum creatinine ≥ 1.1 mg/dl for women and ≥ 1.2 mg/dl for men;
* No organ failure at the time of study enrollment;
* Intervention initiation within 48 hours of ICU admission;
* No history of metastatic cancer or end-stage disease;
* No absolute contraindications to enteral nutrition (e.g., persistent ileus, gastrointestinal ischemia, persistent or biliary vomiting, mechanical obstruction);
* No active infections, sepsis, severe sepsis, or septic shock;
* No intolerance to the whey protein supplement used in the current study;
* Not participating in other clinical trials concurrently with this study;
* No clinical conditions with higher or lower protein needs, such as burns, sepsis, cirrhosis, or chronic kidney disease;
* No diabetes with severe complications such as ketoacidosis, hyperosmolar coma, or acidosis.

Exclusion Criteria:

* Unwillingness to continue cooperation during study;
* Discharge or death of the patient earlier than 5 days from the start of the intervention;
* Occurrence of side effects during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with refeeding syndrome | within the first 5-7 days of nutrition delivery
  Refeeding syndrome will be diagnosed based on a decrease in serum levels of electrolytes, including potassium, magnesium, and phosphate, within the first 5 days of nutrition delivery.

SECONDARY OUTCOMES:
Incidence of infection | Within 5-14 days of nutrition delivery
  Determining and comparing the incidence of infection and its duration
Number of participants with organ failure as measured by SOFA score | Within 5-14 days of nutrition delivery
  Organ failure will be assessed using the SOFA Score (Sequential Organ Failure Assessment), which evaluates the function of the following organ systems:
  Cardiovascular Respiratory Renal Hepatic Coagulation Neurological
Duration of ICU stay | up to 7 weeks after admission
Duration of hospital stay | up to 7 weeks after admission
Mortality | up to 45-day
  45-day mortality from the time of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Vahdat Shariatpanahi Professor, Principal Investigator — School of Nutrition Sciences and Food Technology, Shahid Beheshti University of Medical Sciences
Locations (1):
- Ayatollah Taleghani Medical, Educational, and Therapeutic Center, Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided